CLINICAL TRIAL: NCT04962165
Title: Obstructive Sleep Apnea Management in People With Spinal Cord Injury, Treatment Options by Mandibular Advancement Device
Brief Title: Obstructive Sleep Apnea Management in People With Spinal Cord Injury
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Motol (Other)
Responsible Party: Principal Investigator, Assoc. Prof. Jiri Kriz, MD, PhD, Clinical Professor, University Hospital, Motol
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCI_APNEA_2021
Record Dates: First submitted 2021-01-07; First posted 2021-07-14 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: Obstructive Sleep Apnea; Spinal Cord Injuries
Keywords: Apnea; Spinal cord injury; Mandibular Advancement Device
MeSH Terms: conditions — Sleep Apnea, Obstructive; Spinal Cord Injuries; Apnea | interventions — Occlusal Splints

STUDY DESIGN:
Intervention Model Description: Single Group Assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental group (Experimental): The group of SCI people will use a mandibular advancement device for treatment of obstructive sleep apnea.
  Interventions: Device: Mandibular Advancement Device

INTERVENTIONS:
Device: Mandibular Advancement Device — The device maintain opened upper airway by moving the lower jaw slightly forward while sleeping.

SUMMARY:
The prevalence of obstructive sleep apnea (OSA) is a significantly higher in people after spinal cord injury (SCI) than in the general population. As a positive pressure therapy (CPAP) is often poorly tolerated, a mandibular advancement device (MAD) can be used for the treatment of OSA. The purpose of this study is to determine the efficacy of MAD in people with SCI and to verify their adherence to the therapy.

DETAILED DESCRIPTION:
Obstructive sleep apnea (OSA) is a disorder with serious health consequences. Compared to the general population, a significantly higher prevalence of OSA was found in individuals with spinal cord injury (SCI). As treatment, positive pressure therapy in the respiratory tract during sleep (CPAP) is commonly instituted. However, CPAP therapy is often rejected or poorly tolerated by patients. Alternatively, the American Association of Sleep Medicine recommends the use of Mandibular Advancement Devices (MAD). The MAD prevents the upper airway from collapsing by anterior displacement of the mandible.

The aim of the project is to determine the efficacy of MAD therapy in people with SCI and to verify their adherence to the therapy. The research group will consist of 60-80 subjects. The selection of suitable participants will be based on the results of a polygram. The MAD for a group of subjects with an apnea-hypopnea index (AHI) higher than five will be fabricated using their dental impressions. Subsequently, the subjects will be retested while wearing the MAD and outcomes will be compared. The evaluation will include a set of questionnaires. Adherence to therapy will be checked after three and six months.

The investigators anticipate that the results of the study will confirm the effectiveness of MAD devices in the treatment of OSA in the monitored group. Most importantly, the investigators intend to set a standard for a long-term system of diagnosing and addressing OSA in individuals with SCI.

ELIGIBILITY:
Inclusion Criteria:

* AHI > 5 on polygraphy
* sufficient set of teeth to hold a splint
* written informed consent

Exclusion Criteria:

* use of medication that could affect breathing or sleep
* oxygen-dependent or decompensated lung disease
* decompensated congestive heart failure
* evidence of other sleep disorders (narcolepsy, restless legs syndrome, insomnia)
* abnormalities of the upper airway
* periodontal problems and untreated caries
* mental disorders

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-08-01 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-11-30 (Estimated)

PRIMARY OUTCOMES:
Apnea-Hypopnea index (AHI) | through study completion, an average of 6 month
  The obstructive Apnea-Hypopnea Index is defined as the mean number of obstructive apneas and hypopneas per hour of sleep, thus: the occurrence of 5 to 14 events per hour of sleep means presence of mild apnea, 15 to 29 moderate apnea and ≥ 30 severe apnea. The AHI is derived from overnight polygraphy.

SECONDARY OUTCOMES:
Daytime sleepiness | through study completion, an average of 6 month
  The Epworth sleepiness scale (ESS) will measure the subjective daytime sleepiness, assesses the propensity to sleep under inappropriate circumstances. The ESS questionnaire consists of 8 questions about daytime sleepiness in various situations. The minimum scale values of 0-7 indicate no likeliness of being abnormally sleepy, the maximum scale values of 16-24 indicate excessive sleepiness.
Quality of life measurement | through study completion, an average of 6 month
  The WHOQOL-BREF will be used to measure the quality of life. This instrument is a self-administered questionnaire comprising 26 questions on the individual's perceptions of their health and well-being over the previous two weeks. Scores range from 0 to 100 with 100 indicating a higher quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Jiri Kriz, MD, PhD, Study Director — Spinal Cord Unit, University Hospital Motol
Locations (1):
- Paraple Center - rehab center for SCI people, Prague, Czechia

REFERENCES:
- [Background] Dieltjens M, Vanderveken O. Oral Appliances in Obstructive Sleep Apnea. Healthcare (Basel). 2019 Nov 8;7(4):141. doi: 10.3390/healthcare7040141. PMID 31717429
- [Background] Graco M, Schembri R, Cross S, Thiyagarajan C, Shafazand S, Ayas NT, Nash MS, Vu VH, Ruehland WR, Chai-Coetzer CL, Rochford P, Churchward T, Green SE, Berlowitz DJ. Diagnostic accuracy of a two-stage model for detecting obstructive sleep apnoea in chronic tetraplegia. Thorax. 2018 Sep;73(9):864-871. doi: 10.1136/thoraxjnl-2017-211131. Epub 2018 May 7. PMID 29735608
- [Background] Kriz J., Kyselova A., Sever D. Sleep Apnea In Patients With Chronic Spinal Cord Injury. Abstractbook. The 4th ISCoS and ASIA Joint Scientific Meeting, May 14-16, 2015, Montreal, Canada.